CLINICAL TRIAL: NCT06575985
Title: Investigating the Effects of a 10-day Heat Acclimation and Exercise Intervention on Physiological Adaptations and Cross-tolerance in Women
Brief Title: Mechanisms Underlying Hypoxic, Heat and Cross-tolerance Adaptation in Women
Acronym: FemAdapt_HOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jozef Stefan Institute (Other)
Collaborators: University of Ljubljana (Other); University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Tadej Debevec, Professor, Jozef Stefan Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FemAdapt_HEAT; J5-50180 (Other Grant/Funding Number: Javna Agencija za Raziskovalno Dejavnost RS)
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Heat Exposure; Exercise Training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Considering that the heat acclimation condition will be easily perceptible to the participants, it will not be possible to blind them from their group assignment. The investigators will also be required to set the environmental conditions for each exercise session, so they will also be aware of group assignment during the intervention. However, efforts will be made to blind outcomes assessors to group assignment, by reassigning unique participant identifier codes with the random assignment of "A" and "B" to the experimental and control groups by a third party. The experimental and control group can therefore be compared, without knowledge of which label corresponds to which group until after data processing and statistical analyses have been performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat acclimation and exercise group (Experimental): Experimental group who will complete an exercise training intervention under hot conditions
  Interventions: Other: Heat acclimation and exercise training
- Thermo-neutral exercise training group (Active Comparator): Control group who will complete an exercise training intervention under thermo-neutral conditions
  Interventions: Other: Thermo-neutral exercise training group

INTERVENTIONS:
Other: Heat acclimation and exercise training — 10-day intervention consisting of daily 60-min exercise sessions aimed to induce increases in core body temperature, conducted in a climactic chamber set to 35°C and 50% relative humidity.
  Arms: Heat acclimation and exercise group
Other: Thermo-neutral exercise training group — 10-day intervention consisting of daily 60-min exercise sessions conducted in a climactic chamber set to 23°C and 50% relative humidity.
  Arms: Thermo-neutral exercise training group

SUMMARY:
This study will consist of a parallel-groups design, with 30 healthy active female participants randomly assigned to either an experimental heat acclimation and exercise intervention, or a thermo-neutral exercise intervention control group. Interventions will be 10 days in duration, and consist of daily 60-minute exercise bouts under the appropriate environmental condition. Before and after each intervention, various tests will be conducted to establish exercise capacity under various environmental conditions, as well as underlying mechanisms of physiological adaptation induced by each intervention.

DETAILED DESCRIPTION:
Most research on how the human body responds to different environmental conditions has primarily focused on men, leaving a gap in our understanding of how women adapt to these conditions. Heat exposure in particular is known to affect the well-being and performance of humans, as well as induce chronic adaptations through an acclimation/acclimatization process, which helps the body to better regulate core temperature. Moreover, contemporary research is beginning to explore the 'cross-tolerance' phenomenon; the notion that exposure (and acclimation/acclimatization) to one environmental stressor may affect the responses to another. In particular, both heat and hypoxia are known to activate common acclimatization pathways, with pulmonary, cardiovascular, hematological and muscular adaptations occurring to facilitate both oxygen transport and core body temperature regulation. In line with this background, the primary aim of this study is to investigate the effects of a heat acclimation and exercise intervention, relative to a thermo-neutral exercise control intervention, on exercise tolerance under various environmental conditions (heat, hypoxia, neutral) in healthy, active women. The secondary aim is to establish mechanisms of adaptation, by exploring the intervention-induced changes in pulmonary, cardiovascular, hematological and muscular factors, through various tests conducted at rest and during exercise.

To address these aims, 30 healthy active female participants, aged between 18 and 35 years, will be randomized to either an experimental (heat acclimation and exercise training) or control (thermo-neutral exercise training) group. The experimental group will complete a 10-day heat acclimation training intervention, exercising for 60 minutes per day in a climactic chamber set to 35°C and 50% relative humidity. The control group will complete a similar exercise intervention, but under thermo-neutral conditions (23°C and 50% relative humidity). Before and after the intervention period, both groups will complete a wide variety of tests, including exercise capacity measurements under each environmental condition (heat [35°C], hypoxia [Fraction of inspired oxygen = 0.135], neutral [23°C, FiO2 = 0.209]), body composition assessments, lung function testing, hemoglobin mass and blood volume quantification, skeletal muscle mitochondrial function and vascular responsiveness assessment, and venous blood sampling for a variety of sex hormone-, redox balance-, hematopoietic-, heat shock protein-, hypoxia-inducible factor- and genetic-related markers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 35 years
* Body mass index: 18.5 - 25.0 kg/m^2
* Regular physical activity (at least 30 minutes of moderate-intensity activity, three times per week)

Exclusion Criteria:

* Habitual smoker within the past 5 years
* History of metabolic disorders or any medications deemed to pose an undue risk or introduce bias in any outcome measures
* Exposure to altitude > 2000 m above sea level within four weeks of scheduled participation
* Permanent residence at altitude > 1000 m above sea level

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants will be recruited based on their self-identification as female. Sex hormone measurements will later be conducted to verify alignment between their gender identity and biological sex.
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity under thermo-neutral normoxic conditions | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Results of an incremental exercise test to exhaustion conducted at 23°C and an FiO2 of 0.209, quantified using maximal oxygen uptake
Exercise capacity under hot normoxic conditions | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Results of an incremental exercise test to exhaustion conducted at 35°C and an FiO2 of 0.209, quantified using maximal oxygen uptake
Exercise capacity under thermo-neutral hypoxic conditions | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Results of an incremental exercise test to exhaustion conducted at 23°C and an FiO2 of 0.135, quantified using maximal oxygen uptake

SECONDARY OUTCOMES:
Core body temperature regulation during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Core body temperature measured throughout the incremental exercise tests using a rectal temperature probe.
Skin temperature regulation during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Skin temperature measured throughout the incremental exercise tests using temperature probes attached to the calf, thigh, chest and arm, from which weighted averages are calculated.
Sweat rates during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Sweat rate measured throughout the incremental exercise tests using a sensor attached to the forehead.
Hemo-dynamic activity during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Cardiac output measured throughout the incremental exercise tests by bio-electrical impedance cardiography.
Pulmonary ventilation during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Pulmonary ventilation measured throughout the incremental exercise tests using flow measurements as recorded by metabolic cart.
Gas exchange during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Balance of oxygen uptake and carbon dioxide production measured throughout the incremental exercise tests using gas composition sensors recorded by metabolic cart.
Muscle oxygenation during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Vastus lateralis oxygenation measured throughout the incremental exercise tests using near-infrared spectroscopy.
Brain oxygenation during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Cerebral oxygenation measured at the left pre-frontal cortex throughout the incremental exercise tests using near-infrared spectroscopy.
Pulse oxygen saturation during exercise | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Capillary oxygen saturation measured on the right earlobe throughout the incremental exercise tests using pulse oximetry.
Body composition | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Body mass measured using standard weighing scales, with body fat percentage estimated using a standardized eight-site skinfold measurement protocol with associated equation.
Lung function | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Standard spirometry procedure to assess lung function using forced expiratory volume
Hemoglobin mass | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Hemoglobin mass estimation using the carbon monoxide re-breathing method
Blood/plasma volume | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Blood/plasma volume estimation using the carbon monoxide re-breathing method
Skeletal muscle mitochondrial function | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Skeletal muscle mitochondrial function quantified using a peripheral vascular occlusion test, with the rate of decrease in muscle oxygenation used to estimate mitochondrial function.
Skeletal muscle vascular responsiveness | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Skeletal muscle vascular responsiveness quantified using a peripheral vascular occlusion test, with the rate of increase in muscle oxygenation during re-perfusion, and the oxygenation overshoot relative to pre-occlusion baseline, used to estimate vascular responsiveness.
Blood viscosity | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Blood viscosity will be measured by obtaining venous blood samples from the participants, extracting plasma, and using a cone/plate viscometer to quantify viscosity and varying shear rates.
Oxidative stress marker | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Venous blood samples will be obtained to quantify redox balance from the extracted plasma.
Hematopoiesis | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Venous blood samples will be obtained to measure various markers of hematopoiesis from the extracted plasma, serum and/or whole blood.
Heat shock proteins | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Venous blood samples will be obtained to measure heat shock proteins in the extracted plasma and serum.
Hypoxia-inducible factor 1α | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Venous blood samples will be obtained to measure hypoxia-inducible factor 1α in the extracted plasma and serum.

OTHER OUTCOMES:
Oestrogen | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Oestrogen will be quantified in the plasma extracted from venous blood samples, to identify the menstrual cycle phases of the participants.
Progesterone | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Progesterone will be quantified in the plasma extracted from venous blood samples, to identify the menstrual cycle phases of the participants.
Single nucleotide polymorphisms | Measured once before (pre) and once up to 1 week after (post) the intervention period
  Venous blood samples will be processed and analysed to identify single nucleotide polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Debevec, PhD, Principal Investigator — University of Ljubljana
Locations (2):
- Slovenia (2):
  - Jozef Stefan Institute, Ljubljana, SI
  - University of Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the study, after de-identification, will be made publicly available using an online data repository.
Time Frame: Data will be made available immediately following publication with no end date.
Access Criteria: Any purpose.